CLINICAL TRIAL: NCT04350593
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study Evaluating the Efficacy and Safety of Dapagliflozin in Respiratory Failure in Patients With COVID-19
Brief Title: Dapagliflozin in Respiratory Failure in Patients With COVID-19
Acronym: DARE-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: St. Luke's Hospital, Kansas City, Missouri (Other); AstraZeneca (Industry); Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00081; ESR-20-20653 (Other Grant/Funding Number: Astra Zeneca)
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: sodium-glucose cotransporter-2 inhibitor (SGLT2i); dapagliflozin; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10mg (Active Comparator): Dapagliflozin 10 mg daily
  Interventions: Drug: Dapagliflozin 10 milligram (mg)
- Placebo (Placebo Comparator): Dapagliflozin matching placebo 10 mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 milligram (mg) — Active Comparator: Dapagliflozin 10 mg
  Other Names: Farxiga
  Arms: Dapagliflozin 10mg
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This is an international, multicenter, parallel-group, randomized, double-blind, placebo controlled, study in hospitalized adult patients with coronavirus disease 2019 (COVID-19) in the United States, Brazil, Mexico, Argentina, India, Canada, and United Kingdom. The study is evaluating the effect of dapagliflozin 10 milligrams versus placebo, given once daily for 30 days in addition to background local standard of care therapy, on reducing complications and all-cause mortality, or improving clinical recovery.

DETAILED DESCRIPTION:
COVID-19 can lead to multiorgan failure, especially in high-risk patients. Dapagliflozin, a sodium-glucose cotransporter-2 inhibitor (SGLT2i), favorably impacts many processes dysregulated during acute illness such as COVID-19, has significant cardio- and reno-protective benefits in cardiometabolic disease, and may provide similar organ protection in COVID-19.

The study population will include hospitalized patients with respiratory manifestations of COVID-19 of any duration, but without the need for mechanical ventilation. The eligible patients should have risk factors for developing serious complications of COVID-19, including hypertension, Type 2 diabetes, atherosclerotic cardiovascular disease, heart failure and/or chronic kidney disease stage 3 to 4.

Patients will be treated for 30 days, with either dapagliflozin 10 milligrams daily or placebo, each to be given in addition to the usual standard of care in the participating hospital.

The study assessments include only those that are absolutely critical for ensuring the safety of the patients, to measure efficacy outcomes, and collect biomarker data, so as not to place too high a burden on the study personnel and to minimize additional risk of exposure to severe acute respiratory syndrome coronavirus 2 (SARS CoV-2).

The dual primary efficacy endpoints of the study are time to first event of either complications or death from any cause, and improved clinical recovery through 30 days of follow-up. An extended follow-up period of 60 days (after the 30-day treatment period) is included, in order to examine longer-term trajectory of recovery from COVID-19 among trial participants.

The safety data will be monitored by an Independent Data and Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Male or female patients aged ≥18 years
3. Currently hospitalized
4. Hospital admission no more than 4 days prior to screening
5. Confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by laboratory testing within 10 days prior to screening, or strongly suspected SARS-CoV-2 infection on presentation
6. Chest radiography or computerized tomography (CT) findings that, in the opinion of the investigator, are consistent with coronavirus disease 2019 (COVID-19)
7. Blood oxygen saturation (SpO2) ≥ 94% while receiving low-flow supplemental oxygen (5 liters or less)
8. Medical history of at least one of the following:

   1. hypertension
   2. type 2 diabetes
   3. atherosclerotic cardiovascular disease
   4. heart failure (with either reduced or preserved left ventricular ejection fraction (LVEF))
   5. chronic kidney disease stage 3 to 4 (estimated glomerular filtration rate (eGFR) between 25 to 60 mL/min/1.73 m2)

Key Exclusion Criteria:

1. Respiratory decompensation requiring mechanical ventilation (includes invasive or non invasive ventilation, continuous positive airway pressure (CPAP), or bilevel positive airway pressure (BiPAP))
2. Expected need for mechanical ventilation (includes invasive or non-invasive ventilation, CPAP, or BiPAP) within the next 24 hours
3. Expected survival of less than 24 hours at the time of presentation, in the judgement of the investigator
4. eGFR <25 mL/min/1.73 m2 or receiving renal replacement therapy/dialysis
5. Systolic blood pressure <95 mmHg and/or requirement for vasopressor treatment and/or inotropic or mechanical circulatory support at Screening
6. History of type 1 diabetes mellitus
7. History of diabetic ketoacidosis
8. Currently receiving or has received in the last 14 days, experimental immune modulators and/or monoclonal antibody therapies for COVID-19
9. Current treatment with any sodium-glucose cotransporter-2 inhibitor (SGLT2i) (eg, dapagliflozin, canagliflozin, empagliflozin, ertugliflozin) or having received treatment with any SGLT2i within 4 weeks prior to screening
10. Current participation in another interventional clinical trial (with an investigational drug) that is not an observational registry

    * Note that use of rescue therapies including immune modulators, monoclonal antibody therapies, antiviral therapies, and other agents that are approved or being used through open-label compassionate/expanded use programs or in accordance with the local standard of care is permitted during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kosiborod, MD, Study Chair — Saint Luke's Mid America Heart Institute
Locations (95):
- United States (22):
  - Heart Group of the Eastern Shore, Fairhope, Alabama
  - Baptist Hospital of Miami, Miami, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University, Maywood, Illinois
  - Ascension - St. Vincent, Indianapolis, Indiana
  - Lahey Health, Burlington, Massachusetts
  - McLaren Health Care, Auburn Hills, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - St. Francis Hospital, Roslyn, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Trials Network of Tennessee, Memphis, Tennessee
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - Baylor College of Medicine, Houston, Texas
  - Sentara Healthcare, Norfolk, Virginia
- Argentina (11):
  - Clínica de Especialidades Villa María, Villa María, Province of Córdoba
  - Fundación Favaloro, Buenos Aires
  - Hospital Español, Buenos Aires
  - Hospital Fernández, Buenos Aires
  - Hospital Pirovano, Buenos Aires
  - Hospital Santojanni, Buenos Aires
  - Sanatorio Anchorena, Buenos Aires
  - Sanatorio Güemes, Buenos Aires
  - Clínica Vélez Sarsfield, Córdoba
  - Hospital San Roque, Córdoba
  - Sanatorio Privado Duarte Quiros de Clinica Colombo S.A., Córdoba
- Brazil (35):
  - Centro de Pesquisa Dr. Marco Mota, Maceió, Alagoas
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Unimed de Fortaleza, Fortaleza, Ceará
  - Hospital de Messejana Dr Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - Hospital Estadual Jayme dos Santos Neves, Serra, Espírito Santo
  - Hospital EMEC e Hospital da Cidade, Feira de Santana, Estado de Bahia
  - Hospital e Clínica São Roque, Ipiaú, Estado de Bahia
  - Hospital Regional Deputado Luis Eduardo Magalhães, Porto Seguro, Estado de Bahia
  - Hospital Cárdio Pulmonar, Salvador, Estado de Bahia
  - Hospital Coração do Brasil, Brasília, Federal District
  - Liga de Hipertensão Arterial, Goiânia, Goiás
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital São Domingos - Unimed Uberaba, Uberaba, Minas Gerais
  - PROCAPE, Recife, Pernambuco
  - Hospital Giselda Trigueiro, Natal, Rio Grande do Norte
  - Associação Dr. Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital São José - Criciúma, Criciúma, Santa Catarina
  - IPEMI- Instituto de Pesquisas Médicas de Itajaí, Itajaí, Santa Catarina
  - Hospital Municipal São José, Joinville, Santa Catarina
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Faculdade de Medicina de Botucatu, UNESP, Botucatu, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Unimed Ribeirao Preto, Ribeirão Preto, São Paulo
  - Fundação do ABC (Hospital Estadual Mário Covas), Santo André, São Paulo
  - Centro Integrado de Pesquisas, São José do Rio Preto, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Fundação Pio XII, Barretos
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - Hospital Moriah, São Paulo
  - Hospital Santa Paula, São Paulo
  - InCor - Instituto do Coração do Hospital das Clínicas FMUSP, São Paulo
- Canada (2):
  - Halton Healthcare Services, Oakville, Ontario
  - Lakeridge Health, Oshawa, Ontario
- India (8):
  - CIMS Hospital Pvt. Ltd, Sola, Ahmedabad
  - MIOT International Hospitals, Manapakkam, Chennai-89
  - Sanjivani Super Speciality Hospital Pvt Ltd, Ahmedabad, Gujarat
  - Lokmanya Tilak General Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Science, New Delhi, National Capital Territory of Delhi
  - Max Smart Super Speciality Hospital, Saket, New Delhi
  - Max Super Speciality Hospital (A unit of Devki Devi Foundation), Saket, New Delhi
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
- Mexico (16):
  - Hospital del Prado, Acapulco
  - Icaro Investigaciones en Medicina, Chihuahua City
  - HG de Cuernavaca Dr. Jose G Parres, Cuernavaca
  - JM Research, Cuernavaca
  - Instituto de Investigaciones Aplicadas a la Neurosciencias, Durango
  - Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcade", Guadalajara
  - Hospital San Javier, Guadalajara
  - Invesclinic MX, Guanajuato City
  - CIMEZAP, Jalisco
  - Hospital Medica Sur, Mexico City
  - Hospital Clinica Nova, Monterrey
  - Hospital San Jose TEC Salud, Monterrey
  - ECI Estudios Clinicos Internacionales, Puebla City
  - Hospital SMIQ, Querétaro
  - Investigacion Medica Sonora, Sonora
  - Sanatorio Santa Cruz de Toluca, Toluca
- Addenbrooke's Hospital, Cambridge, CB2 0QQ, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel Jawad M, Furtado RHM, Esterline R, Oscarsson J, Gasparyan SB, Koch GG, Martinez F, Mukhtar O, Verma S, Langkilde AM, Ambery P, Patel S, Gosch K, Windsor SL, Soares RVP, Moia DDF, Aboudara M, Javaheri A, Saraiva JFK, Maia LN, Berwanger O, Sauer AJ, Kosiborod MN. Efficacy and safety of dapagliflozin in patients hospitalized with COVID-19 with and without type 2 diabetes: a prespecified analysis of the DARE-19 randomized trial. Cardiovasc Diabetol. 2025 Jul 30;24(1):307. doi: 10.1186/s12933-025-02875-6. PMID 40739638
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Gasparyan SB, Buenconsejo J, Kowalewski EK, Oscarsson J, Bengtsson OF, Esterline R, Koch GG, Berwanger O, Kosiborod MN. Design and Analysis of Studies Based on Hierarchical Composite Endpoints: Insights from the DARE-19 Trial. Ther Innov Regul Sci. 2022 Sep;56(5):785-794. doi: 10.1007/s43441-022-00420-1. Epub 2022 Jun 14. PMID 35699910
- [Derived] Kosiborod MN, Esterline R, Furtado RHM, Oscarsson J, Gasparyan SB, Koch GG, Martinez F, Mukhtar O, Verma S, Chopra V, Buenconsejo J, Langkilde AM, Ambery P, Tang F, Gosch K, Windsor SL, Akin EE, Soares RVP, Moia DDF, Aboudara M, Hoffmann Filho CR, Feitosa ADM, Fonseca A, Garla V, Gordon RA, Javaheri A, Jaeger CP, Leaes PE, Nassif M, Pursley M, Silveira FS, Barroso WKS, Lazcano Soto JR, Nigro Maia L, Berwanger O. Dapagliflozin in patients with cardiometabolic risk factors hospitalised with COVID-19 (DARE-19): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2021 Sep;9(9):586-594. doi: 10.1016/S2213-8587(21)00180-7. Epub 2021 Jul 21. PMID 34302745

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin 10mg: Dapagliflozin 10 mg daily
  Dapagliflozin 10 MG: Active Comparator: Dapagliflozin 10mg
Period: Overall Study
Arm/Group | Dapagliflozin 10mg | Placebo
Started | 625 | 625
Completed | 617 | 620
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg | Placebo | Total
Number analyzed (Participants) | 625 | 625 | 1250
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.4) | 61.8 (13.5) | 61.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 273 | 533
  Male | 365 | 352 | 717
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: N numbers might differ for some parameters based on data availability.
  Participants
    number analyzed (Participants) | 621 | 619 | 1240
    Hispanic or Latino | 394 | 362 | 756
    Not Hispanic or Latino | 166 | 177 | 343
    Unknown or Not Reported | 61 | 80 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: N numbers might differ for some parameters based on data availability.
  Participants
    number analyzed (Participants) | 623 | 618 | 1241
    American Indian or Alaska Native | 7 | 10 | 17
    Asian | 35 | 29 | 64
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 85 | 84 | 169
    White | 452 | 459 | 911
    More than one race | 43 | 36 | 79
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4
  Argentina | 13 | 14 | 27
  United States | 143 | 144 | 287
  Brazil | 382 | 380 | 762
  United Kingdom | 0 | 2 | 2
  Mexico | 59 | 59 | 118
  India | 26 | 24 | 50
Type 2 diabetes [Count of Participants; unit: Participants] | 312 | 324 | 636
Heart failure [Count of Participants; unit: Participants] | 44 | 46 | 90
Hypertension [Count of Participants; unit: Participants] | 526 | 534 | 1060
Atherosclerotic cardiovascular disease [Count of Participants; unit: Participants] | 93 | 106 | 199
Chronic kidney disease, estimated glomerular filtration rate (eGFR) 25-60 mL/min per 1.73 m^2 [Count of Participants; unit: Participants] | 38 | 44 | 82
Patients with two or more inclusion risk factors [Count of Participants; unit: Participants] | 292 | 319 | 611
Age >/= 60 years [Count of Participants; unit: Participants] | 339 | 360 | 699
Body Mass Index >/= 30 [Count of Participants; unit: Participants] | 296 | 305 | 601
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 25 | 32 | 57
Current smoker [Count of Participants; unit: Participants] | 29 | 20 | 49
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 79.3 (13.7) | 79.7 (13.7) | 79.5 (13.7)
Blood pressure - systolic [Mean (Standard Deviation); unit: mm Hg] | 126.6 (16.0) | 127.0 (16.3) | 126.8 (16.1)
Blood pressure - diastolic [Mean (Standard Deviation); unit: mm Hg] | 76.6 (10.9) | 76.2 (10.6) | 76.4 (10.7)
Temperature [Mean (Standard Deviation); unit: degrees Celcius] | 36.4 (0.6) | 36.4 (0.7) | 36.4 (0.6)
Oxygen saturation [Mean (Standard Deviation); unit: % (measured on supplemental oxygen)] | 95.5 (1.7) | 95.2 (1.8) | 95.3 (1.8)
eGFR [Mean (Standard Deviation); unit: mL/min per 1.73 m^2] | 84.1 (25.0) | 83.4 (24.6) | 83.8 (24.8)
SARS-CoV-2 test result at baseline [Count of Participants; unit: Participants]
  Positive | 584 | 575 | 1159
  Negative | 30 | 35 | 65
  Test results not known | 11 | 15 | 26
Angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) [Count of Participants; unit: Participants] | 225 | 219 | 444
Beta-blocker [Count of Participants; unit: Participants] | 93 | 98 | 191
Calcium blocker [Count of Participants; unit: Participants] | 84 | 88 | 172
Loop-diuretic [Count of Participants; unit: Participants] | 49 | 63 | 112
Statin [Count of Participants; unit: Participants] | 122 | 144 | 266
Anti-coagulant [Count of Participants; unit: Participants] | 527 | 527 | 1054
Biguanide [Count of Participants; unit: Participants] | 82 | 75 | 157
Sulfonylurea [Count of Participants; unit: Participants] | 24 | 22 | 46
Dipeptidyl peptidase 4 (DPP-4) inhibitor [Count of Participants; unit: Participants] | 17 | 11 | 28
Glucagon-like peptide 1 (GLP-1) receptor agonist [Count of Participants; unit: Participants] | 6 | 8 | 14
Insulin [Count of Participants; unit: Participants] | 223 | 221 | 444
Remdesivir [Count of Participants; unit: Participants] | 114 | 111 | 225
Systemic corticosteroids [Count of Participants; unit: Participants] | 176 | 179 | 355
Dexamethasone [Count of Participants; unit: Participants] | 133 | 136 | 269
Other systemic glucocorticoid [Count of Participants; unit: Participants] | 50 | 55 | 105

OUTCOME MEASURES:

1. Primary Outcome: Prevention of COVID-19 Complications or Death: During the 30-day Treatment Period, Time to First Occurrence of New/Worsened Organ Dysfunction During Index Hospitalization or Death From Any Cause.
Description: Time to first occurrence of new/worsened organ dysfunction during index hospitalization or death from any cause.
  Event rates are presented as the number of subjects with event per 100 patient month (30 days) of follow-up.
  Unit of Measure: Patients with events per 100 patient-months (pt-mos) at risk.
  New/worsened organ dysfunction is defined as at least one of the following:
  * Respiratory decompensation requiring initiation of mechanical ventilation (includes invasive or non-invasive ventilation, CPAP, or BiPAP), and/or initiation of extracorporeal membrane oxygenation (ECMO)
  * New or worsening congestive heart failure
  * Requirement for vasopressor therapy and/or inotropic or mechanical circulatory support
  * Ventricular tachycardia or fibrillation lasting at least 30 seconds and/or associated with hemodynamic instability or pulseless electrical activity, or resuscitated cardiac arrest
  * Doubling of s-Creatinine or initiation of renal replacement therapy
Time Frame: Randomization through Day 30
Measure: Number; unit: Patients with events/100 pt-mos at risk
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
Patients with events/100 pt-mos at risk | 12.4 | 15.6

2. Primary Outcome: Improving Clinical Recovery: Hierarchical Composite Outcome Measure Including Death From Any Cause Through Day 30, New/Worsened Organ Dysfunction, Clinical Status at Day 30 and Hospital Discharge Before Day 30 and Alive at Day 30.
Description: The number of patients experiencing improvement by day 30 compared with baseline (discharged from hospital without a worsening event and alive, or still in hospital without a worsening event and without oxygen support) in the hierarchical composite endpoint analysis.
  Hierarchical composite outcome measure includes:
  * Death from any cause through Day 30
  * New/worsened organ dysfunction
  * Clinical status at Day 30 for patients still hospitalized and without any worsening organ dysfunction
  * Hospital discharge before Day 30 and alive at Day 30
Time Frame: Randomization through Day 30
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
participants | 547 | 532

3. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge (refers to index hospitalization only).
  Median time to hospital discharge is presented in days.
Time Frame: Randomization through Day 30
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
days | 5 [5.0 to 6.0] | 6 [5.0 to 6.0]

4. Secondary Outcome: Total Number of Days Alive and Free From Respiratory Decompensation Requiring Initiation of Mechanical Ventilation (Includes Invasive or Non-invasive Ventilation, CPAP, or BiPAP)
Description: Total number of days alive and free from mechanical ventilation (includes invasive or non-invasive ventilation, CPAP, or BiPAP) is calculated for each patient as total follow-up time (30 days) substracted days in hospital with mechanical ventilation and days dead.
Time Frame: Randomization through Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
days | 27.8 (6.8) | 27.4 (7.4)

5. Secondary Outcome: Total Number of Days Alive, Not in the ICU, and Free From Respiratory Decompensation Requiring Initiation of Mechanical Ventilation (Includes Invasive or Non-invasive Ventilation, CPAP, or BiPAP)
Description: Total number of days alive, not in the ICU and free from mechanical ventilation (includes invasive or non-invasive ventilation, CPAP, or BiPAP) is calculated for each patient as total follow-up time (30 days) substracted days in ICU and days dead.
Time Frame: Randomization through Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
days | 27.5 (7.2) | 27.1 (7.7)

6. Secondary Outcome: Time to Composite of Acute Kidney Injury or Initiation of Renal Replacement Therapy, or Death From Any Cause
Description: Acute kidney injury is defined as an episode of doubling s-creatinine compared to baseline during index hospitalization or SAE. Initiation of renal replacement therapy is defined as initiation of renal replacement therapy during index hospitalization or SAE.
  Event rates are presented as the number of subjects with event per 100 patient month (30 days) of follow-up.
  Unit of Measure: Patients with events per 100 patient-months (pt-mos) at risk.
Time Frame: Randomization through Day 30
Measure: Number; unit: Patients with events/100 pt-mos at risk
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
Patients with events/100 pt-mos at risk | 8.2 | 11.2

7. Secondary Outcome: Time to Death From Any Cause
Description: Time to death from any cause.
  Event rates are presented as the number of subjects with event per 100 patient month (30 days) of follow-up.
  Unit of Measure: Patients with events per 100 patient-months (pt-mos) at risk.
Time Frame: Randomization through Day 30
Measure: Number; unit: Patients with events/100 pt-mos at risk
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 625 | 625
Patients with events/100 pt-mos at risk | 6.8 | 9.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing informed consent through the end of the 30-day treatment period.
Description: All-cause mortality was monitored in the total started population of 1250 patients. Serious adverse events, adverse events resulting in the discontinuation of study drug, and safety events of acute kidney injury and diabetic ketoacidosis were monitored in the safety population defined as patients who received at least one dose of study medication. 613 patients in the dapagliflozin group and 616 patients in the placebo group received at least one dose of study medication.
Arm/Group | Dapagliflozin 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 41/625 | 54/625
Serious Adverse Events (participants affected / at risk) | 70/613 | 87/616
Other Adverse Events (participants affected / at risk) | 2/613 | 2/616
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 10mg (N=613) | Placebo (N=616)
COVID-19 (Infections and infestations) | 5 | 3
Septic Shock (Infections and infestations) | 5 | 6
Severe acute respiratory syndrome (Infections and infestations) | 3 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 4
Device related sepsis (Infections and infestations) | 1 | 0
Emphysematous pyelonephritis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Labyrinthitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 8
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pulmonary sepsis (Infections and infestations) | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Euglycemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Ischemic stroke (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Cerebral disorder (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Presnycope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 3 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1
Hypovolemic shock (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 21 | 32
Renal impairment (Renal and urinary disorders) | 1 | 1
Renal injury (Renal and urinary disorders) | 0 | 2
Asthenia (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 3 | 5
General physical health deterioration (General disorders) | 0 | 1
Blood electrolytes abnormal (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac Disorder (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 10mg (N=613) | Placebo (N=616)
Acute Kidney Injury (Renal and urinary disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication with the exception of requiring the removal of confidential information. The embargo can be extended to 90 days if there would be any patent applications to be filed by the sponsor related to the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04350593/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT04350593/SAP_001.pdf